CLINICAL TRIAL: NCT02565654
Title: Efficacy of Rifaximin for Diarrhea-predominant Irritable Bowel Syndrome With Positive Lactulose Hydrogen Breath Test
Brief Title: Efficacy of Rifaximin to Treat Diarrhea-predominant Irritable Bowel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, XiaojunZhuang, doctor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 0717-201506
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome(IBS); Small intestinal bacterial overgrowth (SIBO); Rifaximin
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Faeces
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rifaximin group: Patients are treated with rifaximin (Alfa Wassermann Pharmaceutical Co., Ltd. Italy) for 14 days at a daily dosage of 1200 mg (400 mg, three times daily)

SUMMARY:
Irritable bowel syndrome (IBS) is a common disease and the pathogenesis of this disease includes central and peripheral mechanisms. In recent years, there were many studies suggesting that microbiota in the intestine may play an important role in the IBS.What's more, small intestinal bacterial overgrowth (SIBO) may be an important pathogenic factor for IBS and the use of antibiotics may be beneficial. Therefore, the investigators intend to explore the efficacy of rifaximin for IBS-D in Chinese population.

DETAILED DESCRIPTION:
Recent evidence suggests that a shift in the host-gut microbial relationship as seen in small intestinal bacterial overgrowth (SIBO) may contribute to the pathogenesis of IBS.Overgrowth of microbiota in the small intestine can cause excessive gas production and malabsorption with a variety of nonspecific symptoms, such as diarrhea, gas bloating, abdominal pain and constipation.Glucose (GBT) and lactulose (LBT) breath test have been proposed as simple, inexpensive and non-invasive diagnostic tools for detecting SIBO with respect to the gold standard (the culture of intestinal aspirates). Many antibiotics have been proposed in the last years for SIBO eradication.Rifaximin is a rifamycin derivative with antibacterial activity caused by inhibition of bacterial synthesis of RNA and which is effective against both gram-positive and -negative bacteria, including aerobes and anaerobes.As <0.1% of its oral dose is absorbed, rifaximin administration is associated to a very low side-effect incidence. However,there are still no effective and reliable treatment for IBS,so we intend to explore the prevalence of SIBO in IBS-D patients and evaluate the efficacy of rifaximin for IBS-D in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-65 yr;
2. IBS-D fulfiling the ROME III criteria;
3. had undergone a colonoscopic examination within the previous 2 years;
4. had received a diagnosis of and had current symptoms of IBS, in particular, symptoms of abdominal pain and discomfort; and did not have adequate relief of global IBS symptoms and of IBS-related bloating at both the time of screening and the time of randomization.

Exclusion Criteria:

1. age <18 years;
2. use of antimicrobial agents within the previous 3 months;
3. known hypersensitivity to agents belonging to rifamycin and/or tetracycline families;
4. pregnancy or breast-feeding;
5. evidence of major concomitant diseases (including tumours and hepatic and ⁄ or renal insufficiency);
6. not on antibiotic treatment or probiotics for at least 4 weeks prior to undergoing the LHBT;
7. fibre supplements or laxatives 1-week prior to the LHBT test date
8. presence of endoscopic or histological alterations, which might be indicative of other disorders (e.g. celiac disease, inflammatory bowel disease, diverticulosis or diverticulitis) and contribute to IBS symptom generation,
9. evidence of major concomitant diseases (including tumours and hepatic and/or renal insufficiency)
10. unstable thyroid disease
11. bowel obstruction
12. known lactose intolerance
13. any evidence of advanced organic or psychiatric disease that may impact on the patient's compliance or adherence to the study protocol.
14. use of medications known to cause constipation (eg, narcotics, antidiarrheals, alosetron)
15. history of abdominal surgery involving the gastrointestinal tract such as appendicectomy, cholecystectomy
16. Inability to sign or rejection to informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 40 cases of LHBT positive and 20 cases of LHBT negative IBS-D patients will be included in this study. The estimate of the LHBT positive rate was 40%, so we need to screen about 100 IBS-D patients. We are going to recruit 120 IBS-D patients in our center with respect to patients lost to follow up.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients who had adequate relief of global IBS symptoms | 12 weeks

SECONDARY OUTCOMES:
the proportion of patients who with positive lactulose hydrogen breath test change to be negative | 2 weeks
the composition of patients's fecal microbiota | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The first Affiliated Hospital of Sun Yat-Sen university, Guangzhou, Guangdong, China